CLINICAL TRIAL: NCT04201028
Title: A Remote Delivered Lifestyle Therapeutics Program: A Randomized Clinical Trial
Brief Title: A Remote Delivered Lifestyle Therapeutics Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coastal Carolina University (Other)
Collaborators: inHealth Medical Services, Inc. (Industry)
Responsible Party: Principal Investigator, Kelly Johnson, Assistant Professor of Exercise and Sport Science, Coastal Carolina University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021.96
Record Dates: First submitted 2019-12-13; First posted 2019-12-16 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Body Weight Changes; Weight Loss; Healthy Diet; Obesity
Keywords: telehealth; video conferencing; blood pressure; lipids; weight loss; usual care; obesity medicine
MeSH Terms: conditions — Body Weight Changes; Weight Loss; Obesity | interventions — Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: All participants were randomized in a balanced fashion and stratified by sex into either one of the two intervention groups no device (NODEV) group or a device (DEV) group.
Who Masked: Care Provider
Masking Description: Following baseline visits, participants were randomized to a no device (NODEV) or device (DEV) group via the website https://www.randomlists.com/team-generator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Conferencing Health Coaching with devices (Experimental): The DEV group participants will meet via the DiscoverHealth® app using their smartphone, and met 18 times with the registered dietitian (RD) to discuss exercise and diet goals. Participants in this group were provided with a blood pressure and body weight scale which connected to the CoachCare App®.
  Interventions: Behavioral: Video Conferencing Health Coaching with devices
- Video Conferencing Health Coaching with no devices (Experimental): The NODEV group participants meet via the DiscoverHealth® app using their smartphone, and met 18 times with the registered dietitian (RD) for health coaching to discuss exercise and diet goals. Participants in this group did not receive devices.
  Interventions: Behavioral: Video Conferencing Health Coaching with no devices

INTERVENTIONS:
Behavioral: Video Conferencing Health Coaching with devices — Devices
  Arms: Video Conferencing Health Coaching with devices
Behavioral: Video Conferencing Health Coaching with no devices — No Devices
  Arms: Video Conferencing Health Coaching with no devices

SUMMARY:
Heart disease is the leading cause of death in the United States. The overall risk for heart disease is a composite measure of various modifiable factors including blood pressure, cholesterol, and tobacco use; which are exacerbated by a sedentary lifestyle, unhealthy diet, and being overweight. Approximately 32% of the adult U.S. population has high blood pressure and 46% of them have uncontrolled hypertension. Successful management of high blood pressure and other cardiovascular risk is a complex process that requires significant lifestyle changes but adopting and adhering to these changes is challenging. A promise approach to overcoming these challenges is utilizing health coaching. The purpose of this research study is to compare at home devices for blood pressure and weight measurements (DEV) group compared to not using any at home devices Group (NODEV). Both groups will be supported throughout this study by meeting with obesity medicine doctor monthly in office and have a virtual health coaching visits throughout the study duration.

DETAILED DESCRIPTION:
Baseline Assessment Participants attend a baseline assessment with a study Health Coach that includes an overview and explanation of the study, the completion of several surveys that involve questions related to your overall health and demographics (age, race, etc). In addition, body weight using a scale and resting blood pressure using a blood pressure cuff. During participants will be asked to download the DiscoverHealth app which will be used to track daily nutritional information (food and drinks) and for health coaching sessions.

Groups Participants will then be randomly assigned to a device group (DEV) or a no device group (NODEV).

Control Group If randomly assigned to the NO DEV Group, participants will be asked to download the DiscoverHealth® app and daily input their nutritional information into the app. This will occur at the baseline assessment. Monthly participants will be asked to attend the Sleep Health Clinic to obtain body weight and blood pressure.

Intervention Group

Regardless of randomization (NODEV OR DEV) participants will be be asked to input their daily nutritional information (food) into the DiscoverHealth® app which will be used by the medical doctor and health coach.

Physical Activity Recommendations:

They will be asked to exercise in accordance with obesity medicine doctors recommendations which may be recommendations like obtaining 20 minutes per day of walking with gradual progression to at least 60 minutes per day and achieve 10,000 steps/day. These recommendations are consistent with the guidelines of national organizations.

No Device Group (NODEV):

Medical Doctor Visits:

If participants are randomized to the NODEV group they will individually meet at the Sleep health Clinic and meet with the obesity medical doctor monthly (1-6) with each visit lasting approximately 15 - 45 minutes per visit. During the first visit each subject will be provided with individualized targets for the number of calories to consume per day and associated macronutrient ratios (i.e. percent of calories from protein, fat, and carbohydrates). They will be asked to follow diet recommendations which emphasizes fruits, vegetables, and low-fat dairy foods and reduced consumption of saturated fat, total fat, and cholesterol along with whole grains, poultry, fish, and nuts. The obesity medicine doctor will prescribe calories. At each visit body weight and blood pressure will be assessed and recorded, and the medical doctor will review and discuss each subject's current diet, physical activity plan, body weight and blood pressure changes.

Health Coaching Visits:

Months 1-3: Following the initial baseline visit they receive weekly individualized video health coaching sessions through the video conference feature of the DiscoverHealth® app on your Apple iPhone® or Android® smart phone. These health coaching sessions will be separate video conferences with the research team's Health Coach (HC). During these sessions, they will receive weekly educational online modules focusing on nutrition and fitness as well as education on way to manage your high blood pressure. Each week, the HC will review their progress including calories per day, macronutrient ratio, and make changes to your meal plan if needed. Additionally, the HC will discuss the physical activity program and progress it as needed (i.e. increase the number of steps per day). Each health coaching session will last approximately 20 minutes each resulting in a time subject commitment of 40 minutes per week. During all sessions, participants will have time to express any concerns or questions you may have.

Months 4-6: All health coaching session information and follow up will remain the with the health coach except participants will receive bi-weekly video health coaching sessions through the video conference feature of the DiscoverHealth® app on your Apple iPhone® or Android® smart phone. They will meet 6 times with the health coach during these months.

Device Group (DEV):

Months 1-3: Following the initial baseline visit participants will receive weekly video health coaching sessions through the video conference feature of the DiscoverHealth® app on their Apple iPhone® or Android® smart phone. These health-coaching sessions will be separate video conferences with the research team's HC. During these sessions, they will receive weekly educational online modules focusing on nutrition, fitness, behavior modification, and support building as well as education on ways to manage their blood pressure. Each week, they will be asked to weigh themselves and take their blood pressure using the devices provided, daily. They will meet with the HC each week to review your progress including calories per day, macronutrient ratio, and make suggestions to their meal plan if needed. Additionally, the HC will discuss the physical activity program and progress it as needed (i.e. increase the number of steps per day). Each health coaching session with HC will last approximately 20 minutes each resulting in a time subject commitment of 40 minutes per week. During all sessions, they will have time to express any concerns or questions you may have. They will meet 12 times with the registered dietitian during these months.

Months 4-6: All health coaching session information and follow up will remain the with the HC except they will receive bi-weekly individualized video health coaching sessions through the video conference feature of the DiscoverHealth® app on their Apple iPhone® or Android® smart phone. Each week, they will still be asked to weigh themselves and take their blood pressure using the devices provided, daily. They will meet 6 times with the health coach and during these months.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English spoken and written at a high-school level, Obese according to body mass index (BMI) standards (> 30 kg/m2), Weigh less than 500 pounds, have access to an Apple® iPhone or Android® smart phone

Exclusion Criteria:

* Participants were excluded if they have stated having an Immunodeficiency disorder Kidney disease; Type II diabetes; Asthma, COPD, Heart attack or stroke within the past 12 months; Presence of a partial or full artificial limb; Known dementia, brain cancer, eating disorders, history of significant neurological or psychiatric disorder or any other psychological condition; Medications, dietary supplements, or substances advertised to modify metabolism or body weight; Undergone major surgery less than 4 weeks prior to enrollment in the study; or were actively losing weight.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-12 (Actual)

PRIMARY OUTCOMES:
Weight loss | Change in weight between baseline (week 0) and post intervention (week 26) ]
  Investigators examined body weight changes between groups baseline (week 0) and post intervention (week 26).
Blood Pressure | Change in blood pressure between baseline (week 0) and post intervention (week 26) ]
  Investigators examined blood pressure changes between groups baseline (week 0) and post intervention (week 26).

SECONDARY OUTCOMES:
HbA1c | Pre and Post (a 26 week study)
  Investigators measured HbA1c via a blood test which was analyzed by Quest® laboratories.
Lipid Panel | Pre and Post (a 26 week study)
  Investigators measured HDLs, LDLs, Cholesterol, and Triglycerides via a blood test which was analyzed by Quest® laboratories.

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Health Clinic, Bradenton, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Svetkey LP, Simons-Morton D, Vollmer WM, Appel LJ, Conlin PR, Ryan DH, Ard J, Kennedy BM. Effects of dietary patterns on blood pressure: subgroup analysis of the Dietary Approaches to Stop Hypertension (DASH) randomized clinical trial. Arch Intern Med. 1999 Feb 8;159(3):285-93. doi: 10.1001/archinte.159.3.285. PMID 9989541
- [Background] Alencar MK, Johnson K, Mullur R, Gray V, Gutierrez E, Korosteleva O. The efficacy of a telemedicine-based weight loss program with video conference health coaching support. J Telemed Telecare. 2019 Apr;25(3):151-157. doi: 10.1177/1357633X17745471. Epub 2017 Dec 3. PMID 29199544
- [Background] Johnson KE, Alencar MK, Coakley KE, Swift DL, Cole NH, Mermier CM, Kravitz L, Amorim FT, Gibson AL. Telemedicine-Based Health Coaching Is Effective for Inducing Weight Loss and Improving Metabolic Markers. Telemed J E Health. 2019 Feb;25(2):85-92. doi: 10.1089/tmj.2018.0002. Epub 2018 May 30. PMID 29847222
- [Background] American Heart Association; American College of Cardiology; Obesity Society. Reprint: 2013 AHA/ACC/TOS Guideline for the Management of Overweight and Obesity in Adults. J Am Pharm Assoc (2003). 2014 Jan-Feb;54(1):e3. doi: 10.1331/japha.2014.14502. No abstract available. PMID 24898716